CLINICAL TRIAL: NCT05664204
Title: Veno-arterial Extracorporeal Membrane Oxygenation to Reduce Morbidity and Mortality Following Lung Transplant: a Randomized Controlled Trial
Brief Title: Veno-arterial ExtraCorporeal Membrane Oxygenation to Reduce Morbidity and Mortality Following Lung TransPlant
Acronym: ECMOToP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: APHP211037; 2022-A00538-35 (Other: ID-RCB)
Record Dates: First submitted 2022-12-07; First posted 2022-12-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: The Number of Ventilator-free Days in the 28 Days Following LT
MeSH Terms: interventions — Extracorporeal Membrane Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Systematic ECMO (Experimental): VA-ECMO will be implanted before the first pulmonary artery cross-clamp, in a systematic manner
  Interventions: Procedure: Veno-arterial extracorporeal membrane oxygenation
- On-demand ECMO (Active Comparator): VA-ECMO will be implanted intraoperatively, in an unplanned manner if the hemodynamic and respiratory indices meet pre-planned criteria at different time-points:
  a PaO2/FiO2 ratio<100 mmHg or a respiratory acidosis, with pH< 7.2, PaCO2>60 mmHg, a mean pulmonary arterial pressure>50mmHg (or 2/3 of MAP) and/or an acute pulmonal core at trans-esophageal echography monitoring an acute left ventricular dysfunction at trans-esophageal echography monitoring
  Interventions: Procedure: Veno-arterial extracorporeal membrane oxygenation

INTERVENTIONS:
Procedure: Veno-arterial extracorporeal membrane oxygenation — Strategy would reduce the need for invasive mechanical ventilation in the first 28 days without increasing adverse events

SUMMARY:
In patients undergoing lung transplantation (LT), the investigators hypothesize that a "systematic" intraoperative ECMO strategy would reduce the need for invasive mechanical ventilation in the first 28 days without increasing adverse events, as compared to an "on-demand" intraoperative ECMO strategy.

To date, LT remains a highly hazardous procedure. Even if the surgical procedure is well established, the intraoperative support is not, and most intra-operative ECMO decisions rely on local protocols, anesthesiologists' habits, and surgeons' preference.

The efficacy of applying a "systematic" strategy on reducing the occurrence of severe primary graft dysfunction and thus mechanical ventilation in the 28 days following LT, without increasing mortality or morbidity, would support future guidelines on the use of ECMO in the intraoperative period of LT for obstructive and restrictive lung diseases.

DETAILED DESCRIPTION:
Lung transplantation (LT) provides the prospect of improved survival and quality of life for patients with end stage lung and pulmonary vascular diseases. Its performance carries significant adverse effects, being either intra- or postoperative. The ventilation of a diseased lung for sometimes extended periods and the risk of reperfusion oedema and primary graft dysfunction is a challenge. Moreover, significant hemodynamic instabilities episodes might occur, because of pressure on, or displacement of the heart, clamping of the pulmonary arteries and ischemia-reperfusion syndrome. veno-arterial extracorporeal membrane oxygenation (VA-ECMO) has now replaced cardiopulmonary bypass for respiratory and hemodynamic intraoperative support, carrying less side effects, and an improved early survival.

Even though ECMO is a widely used technique, no precise guideline exists on the hemodynamic and respiratory indexes in LT settings to initiate intraoperative ECMO, but only experts' opinion. Besides, it has to be underlined that the rate of LT performed in the absence of any mechanical support is highly variable among centres, ranging from being exceptional up to 70%.

The investigators aim at evaluating two strategies of ECMO initiation in the pre- and intraoperative periods in patients with pulmonary disease requiring LT: an "on-demand" strategy, in which VA-ECMO will be initiated on high hemodynamic and respiratory needs thresholds and a "systematic" strategy in which VA-ECMO will be pre-emptively initiated.

The investigators hypothesize that a "systematic" strategy allows to reduce the risk of severe primary graft dysfunction and the need for mechanical ventilator in the 28 days following LT without increasing adverse events

ELIGIBILITY:
Inclusion Criteria:

Age >18 years Assessed for bilateral sequential lung transplantation for obstructive or restrictive lung disease Affiliation to the French social security Written informed consent

Exclusion Criteria:

At listing :

* a pulmonary hypertension with a mPAP > 45 mmHg, including in the absence of haemodynamic collapse (MAP, LVEF, RV function all normal)
* a pulmonary hypertension with echocardiographic evidences of right heart dysfunction (paradoxical septum or RV dilatation or RVEF < 35%)
* a pre-capillary pulmonary hypertension at right heart catheterization with low cardiac output

  * LT for primary pulmonary hypertension
  * LT for cystic fibrosis and graft-vs-host disease
  * Re-do LT
  * Combined multi-organ transplantation
  * Active malignancy
  * Pregnancy, breastfeeding
  * Patients under guardianship (tutelle, curatelle, sauvegarde de justice)

Socondary exclusion criteria:

Patients without pulmonary hypertension or with pulmonary hypertension without right ventricular dilatation on an echocardiography in the last 6 months will be randomized; Patients meeting one of the following criteria will not be randomized and will be secondary excluded from the study :

* preoperative severe pulmonary hypertension with hemodynamic collapse on echocardiography defined by: paradoxical septum or dilatation of the right ventricle or RVEF < 20LT in a patient under ECMO as bridge-to-transplantation
* PreLT hypoxemia with PaO2/FiO2 < 80mmHg
* PreLT hypercapnia PaCO2 > 80 mmHg after induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-09-28 (Estimated)

PRIMARY OUTCOMES:
The number of ventilator-free days | The 28 days following LT
  Assess the efficacy of a systematic, pre-operative VA-ECMO strategy on increasing ventilator-free days in the 28 days following LT

SECONDARY OUTCOMES:
The occurrence of grade III PGD | The 72 hours following LT
All-cause mortality | Day-90 after LT
Vital status | Day-90 after LT
Time-to-death from all causes | The first year after LT
The occurrence of ECMO-associated adverse event ; ECMO-associated adverse event defined as cannula infection, misplacement, intra-operative or per-ECMO air-embolism, limb ischemia, vascular complications, thrombophlebitis | The 28 days following LT, Assessed daily from day-1 to day-90
The occurrence of ventilator associated pneumonia (VAP) ; Occurrence of VAP (microbiologically confirmed pneumonia occurring under invasive ventilation 21 and after 48 hours of invasive ventilation) | The 28 days following LT
The occurrence of intraoperative hemodynamic failure; | The 28 days following LT
  Intra-operative amount of norepinephrine (dose in microg/kg of body weight)
The occurrence of post-operative hemodynamic failure ; | The 28 days following LT
  Norepinephrine-free days (number of days without noradrenaline administration)
The occurrence of acute renal failure; | The 28 days following LT
  Renal failure KDIGO stage 3
The need of red blood cell transfusion | The 28 days following LT
  Number of red blood cell packs administered
ECMO-free days ; VV or VA-ECMO-free days | The 28 days following LT
The length of intensive care unit stay | at day 90
  Length of ICU stay in days
The length of hospital stay; Length of hospital stay in days | at day 90
The occurrence of bronchial complication requiring a bronchoscopic intervention ; Bronchial complications requiring a bronchoscopic intervention | From LT to 1-year
Forced expiratory volume during the first second (FEV1) | At 1-year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan MESSIKA, MD, Principal Investigator — Hôpital FOCH
Locations (2):
- France (2):
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital FOCH, Suresnes

IPD SHARING:
Plan to Share IPD: Yes
participant-level deidentified dataset
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Up to two years after the last publication of the research results
Access Criteria: IPD and any additional supporting information will be available on reasonable request from the corresponding author, for additional analyses such as -but not limited to- metaanalyses. The scientific advisory board of ECMOTOP study will assess the relevance of the request.

REFERENCES:
- [Derived] Messika J, Eloy P, Boulate D, Charvet A, Fessler J, Jougon J, Lacoste P, Mercier O, Portran P, Roze H, Sage E, Thes J, Tronc F, Vourc'h M, Montravers P, Castier Y, Mal H, Mordant P; Investigators from the ECMOToP Study group. Protocol for venoarterial ExtraCorporeal Membrane Oxygenation to reduce morbidity and mortality following bilateral lung TransPlantation: the ECMOToP randomised controlled trial. BMJ Open. 2024 Mar 5;14(3):e077770. doi: 10.1136/bmjopen-2023-077770. PMID 38448059